CLINICAL TRIAL: NCT00246103
Title: Phase I Trial of Valproic Acid and Epirubicin in Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13693; USFIRB#101881
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2009-01

CONDITIONS: Neoplasms, Advanced
Keywords: Valproic Acid; Epirubicin; Solid Tumor; Malignancies
MeSH Terms: conditions — Neoplasms | interventions — Valproic Acid; Epirubicin; Fluorouracil; Cyclophosphamide

ARMS (1):
- Dose Escalation and Possible Expansion (Experimental): Escalating doses of Valproic acid and one dose escalation step of epirubicin. Participants with breast cancer treated at the maximum tolerated dose, will also be treated with 5-fluorouracil and Cyclophosphamide.
  Interventions: Drug: Valproic acid; Drug: Epirubicin; Drug: 5-fluorouracil; Drug: Cyclophosphamide.

INTERVENTIONS:
Drug: Valproic acid — Beginning Dose, Level 1: 15 mg/kg/day.
  Other Names: Valproic; Depakote; VPA
Drug: Epirubicin — Beginning Dose, Level 1: 75 mg/m^2.
  Other Names: Ellence
Drug: 5-fluorouracil — For breast cancer participants treated at MTD of Valproic acid and Epirubicin: 5-fluorouracil 500 mg/m^2.
  Other Names: 5-FU
Drug: Cyclophosphamide. — For breast cancer participants treated at MTD of Valproic acid and Epirubicin: cyclophosphamide 500 mg/m^2.
  Other Names: CYTOXAN®

SUMMARY:
This is a Phase I dose escalation trial with escalating doses of Valproic acid and one dose escalation step of epirubicin. VPA will be escalated starting at a dose that is recommended for use as an anti-convulsant or to treat migraine headaches. Epirubicin will be given by infusion on day 3 after the last dose of divalproex. The study will determine the highest dose that these two drugs can be given together and as part of a multidrug regimen with 5-fluorouracil and cyclophosphamide.

DETAILED DESCRIPTION:
This is a Phase I dose escalation trial with escalating doses of Valproic acid and one dose escalation step of epirubicin. VPA will be escalated starting at a dose that is recommended for use as an anti-convulsant or to treat migraine headaches. Recommended concentrations for seizure control is 15-60 mg/kg. Pharmacokinetic studies from healthy volunteers and patients suggested a linear increase in plasma concentrations. A daily dosing of 16 mg/kg divalproex (delayed-release VPA) resulted in a peak VPA plasma concentration of 127 μg/ml (~0.9 mM) 27. The recommended Phase II dose of VPA was 60 mg/kg/d when given by a one-hour intravenous infusion twice daily for 5 days every three weeks.

Synergistic activity between VPA and epirubicin has been observed at 0.5 mM of VPA in our preclinical laboratory studies. Patients will receive an intravenous loading dose of VPA followed by divalproex in two daily doses for 5 doses. The loading dose of VPA will avoid a delay in peak plasma concentrations and excessive nausea. Epirubicin will be given by infusion on day 3 after the last dose of divalproex.

Once the MTD for this two drug regimen has been determined, the maximum tolerated dose will be determined as part of the FEC regimen (5-fluorouracil, epirubicin and cyclophosphamide).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have cytologically/histologically documented solid tumor malignancies
* Age > 18 years old
* Patients must have ECOG performance status 0-2
* Patients must be able to give informed consent and able to follow guidelines given in the study
* The patient has no major impairment of hematological function, as defined by the following laboratory parameters: WBC >3.0x109/L; ANC > 1.5 x 109/L; Hgb >9.0g/dL; PLT >100x109/L (untransfused). Red blood cell transfusions and repeat evaluations for study entry are allowed
* All patients of reproductive potential must use an effective method of contraception during the study and six months following termination of treatment. (Not applicable to patients with bilateral oophorectomy and/or hysterectomy or to female patients who are older than 50 years and have not had a menstrual cycle in more than one year.
* Patients must have measurable or evaluable disease by staging studies performed within 4 weeks of enrollment (evaluable disease refers to ovarian cancer with an elevated CA-125 or prostate cancer with elevated PSA only)
* Once MTD for VPA and epirubicin is reached, the trial will be limited to patients with breast cancer
* At the MTD for VPA and FEC MTD for the trial will be expanded to 15 patients with advanced (inflammatory, Stage >IIIB or regional stage IV) or metastatic breast cancer.
* Patients must have biopsiable disease and be willing to undergo pre and post-VPA biopsies in cycle 1; Patients must have measurable disease, Patients from the last cohort may be included if they were biopsied

Exclusion Criteria:

* Patients may not have had cumulative anthracycline exposure greater than doxorubicin 300 mg/m2 or epirubicin 600 mg/m2.
* Patients must not have evidence of significant active infection (e.g., pneumonia, cellulitis, wound abscess, etc.) at time of study entry.
* Patients must have adequate renal and normal hepatic function (creatinine < 1.5 x upper limit of normal (ULN), bilirubin and SGOT (AST), SGPT (ALT) within 1.5 x the upper institutional normal limits) obtained within 4 weeks prior to registration.
* Pregnant and breast feeding women are excluded from the study because effects on the fetus are unknown and there may be a risk of increased fetal wastage.
* Women of childbearing age must have a negative pregnancy test and be willing to use a highly effective method of contraception. Men who are sexually active must also be willing to use an accepted and effective method of contraception.
* Patients taking anti-arrhythmic medication or with a history of cardiac failure or with ejection fraction £ 50 % are excluded. Patients with a history of long QT syndrome are excluded from study. Patients with a history of ventricular tachycardia or fibrillation are also excluded. Patients must have normal sinus rhythm and normal PR and QT intervals on EKG.
* Patients with uncontrolled CNS metastasis or a history of seizures are excluded. Patients with stable CNS metastasis (either surgically resected, treated with gamma knife or stable for 3 months following WBRT are eligible)
* Patients with stable brain metastases will need an MRI within 4 weeks prior to start of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2004-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Up to 2 months
  MTD of Valproic acid in combination with Epirubicin. The maximum tolerated dose (MTD) will be defined as the highest dose level at which less than 2 out of 6 patients (<33%) experience DLT in Cycle 1. A dose limiting toxicity (DLT) will be defined as any one of the specific adverse events (AEs) outlined in the protocol, occurring during Cycle 1 when considered related to therapy that is part of this study.

OTHER OUTCOMES:
Pharmacokinetic Profile | 6 months
  To determine the pharmacokinetic profile of valproic acid and epirubicin in this combination.
VPA effects on Histone Acetylation | 6 months
  To determine VPA effects on histone acetylation in peripheral blood mononuclear cells and VPA effects on histone acetylation and epirubicin induced DNA damage in biopsied tumors.
MTD for VPA and Epirubicin in Combination with 5-fluorouracil and Cyclophosphamide | 6 months
  To determine the MTD for VPA and epirubicin in combination with 5-fluorouracil and cyclophosphamide commonly known as a regimen called FEC100.
Utility of Topo IIα and IIβ as Predictive Factors for Response | 6 months
  To determine the utility of topo IIα and IIβ as predictive factors for response and their modulation as drug targets in patients with biopsied tumors and to document any responses to this combination.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Munster, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute; Adil Daud, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States